CLINICAL TRIAL: NCT04335669
Title: A Translational Randomized Phase III Study Exploring the Effect of the Addition of Capecitabine to Carboplatine Based Chemotherapy in Early "Triple Negative" Breast Cancer
Brief Title: NordicTrip, a Translational Study of Preoperative Chemotherapy in TNBC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Collaborators: Swedish Breast Cancer Group (Other); Danish Breast Cancer Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NBG-19-01; SWEBCG 19-01
Record Dates: First submitted 2019-12-02; First posted 2020-04-06 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Triple Negative Breast Neoplasms
Keywords: Breast neoplasms; Triple negative breast neoplasms; Neoadjuvant treatment; Translational research; Pathologic response; Pathologic complete response; epirubicin; cyclophosphamide; paclitaxel; carboplatin; capecitabine; Survival outcomes; Homologous repair deficiency; pembrolizumab
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms; Pathologic Complete Response | interventions — Epirubicin; Cyclophosphamide; Paclitaxel; Carboplatin; pembrolizumab; Anthracyclines; taxane; Platinum; Capecitabine; Antimetabolites

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Platinum-based dose dense EC): (Active Comparator): ddEC x 4 + pembrolizumab→ PK x 4 + pembrolizumab, Two-weekly epirubicin/cyclophosphamide (EC) x 4 (epirubicin 90 mg/m2 and cyclophosphamide 600 mg/m2), followed after a three-week interval by three-weekly carboplatin x 4 (AUC = 5) together with weekly paclitaxel x 12 (80 mg/m2). Pembrolizumab is given as a 400 mg iv dosis every 6 weeks for the duration of preoperative chemotherapy.*
  Interventions: Drug: epirubicin, cyclophosphamide, paclitaxel, carboplatin, pembrolizumab
- Arm B (Platinum-based with capecitabine): (Experimental): CEX x 4→ PK x 4, Three-weekly cyclophosphamide/epirubicin/capecitabine (CEX) (epirubicin 75 mg/m2, cyclophosphamide 600 mg/m2 and capecitabine 900 mg/m2) x 4, followed after a three-week interval by three-weekly carboplatin x 4 (AUC = 5) together with weekly paclitaxel x 12 (80 mg/m2).Pembrolizumab is given as a 400 mg iv dosis every 6 weeks for the duration of preoperative chemotherapy.*
  *The addition of pembrolizumab is strongly recommended to all participating patients. However, patients with a documented contraindication, or unwilling to receive immunotherapy may be included in the study without the administration of pembrolizumab.
  Interventions: Drug: epirubicin, cyclophosphamide, capecitabine, paclitaxel, carboplatin, pembrolizumab

INTERVENTIONS:
Drug: epirubicin, cyclophosphamide, paclitaxel, carboplatin, pembrolizumab — Cytotoxic agents.
  Other Names: anthracycline, taxane, platinum
  Arms: Arm A (Platinum-based dose dense EC):
Drug: epirubicin, cyclophosphamide, capecitabine, paclitaxel, carboplatin, pembrolizumab — Cytotoxic agents.
  Other Names: anthracycline, taxane, antimetabolite, platinum
  Arms: Arm B (Platinum-based with capecitabine):

SUMMARY:
Primary aim: To compare the effect on pathologic complete response (pCR) rate of adding capecitabine to carboplatin based preoperative chemotherapy in early ER-negative and HER2-negative breast cancer. Pembrolizumab is allowed in both arms after approval for TNBC 2022.

DETAILED DESCRIPTION:
Primary aim: Pathological complete response rate after preoperative chemotherapy is the primary end-point of the study, which will be evaluated by comparing the effects of neoadjuvant administration of a carboplatin-based treatment and treatment adding capecitabine on pCR. After the approval of pembrolizumab in the preoperative treatment of early TNBC in 2022 the study will consist of two cohorts, one (cohort 1) without the addition of pembrolizumab, and one (cohort 2) with the addition of pembrolizumab to both study arms. The primary evaluation will be performed on the entire study population including both cohorts.

Primary translational aim: To investigate if the effects of the treatments depend on homologous repair deficiency (HRD)-status. More specifically, the aim is to test for differential effect of the two treatments on pCR for HRD-negative (HRD low and intermediate by oncoscan) and HRD-positive (HRD high by oncoscan) patients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent approved by the Ethical Review Board (IRB).
2. Age ≥ 18 to < 76 years.
3. Histologically confirmed unilateral adenocarcinoma of the breast where neoadjuvant chemotherapy followed by definitive surgery is planned.
4. Node positive disease (N1-3) or if clinically N0 Tumor size >20 mm. When deciding T-stage the following hierarchy applies,

   1. MRI
   2. Ultrasound
   3. Mammography
   4. Clinical examination
5. ER negative tumor defined by at least one the following:

   1. ER < 1% cells positive by immunohistochemistry (IHC) or ER ≤ 10% cells positive by IHC and basal-like subtype using gene expression analysis
   2. ER < 10% cells positive by IHC and PgR < 10% cells positive by IHC
6. HER2-normal tumor defined according to applicable national guidelines
7. Consent for germline mutation screening for BRCA1, BRCA2 and other inherited breast cancer associated genes.
8. WHO performance status 0 or 1.
9. Negative pregnancy test in women of childbearing potential (premenopausal or <12 months of amenorrhea post-menopause and who have not undergone surgical sterilization).
10. Willingness of female patients of childbearing potential, male patients, and their sexual partners to use an effective means of contraception during the treatment period and at least 6 months thereafter.
11. Willingness by the patient to undergo treatment and study related procedures according to the protocol.

Exclusion Criteria:

1. Clinical or radiological signs of metastatic disease.
2. History of other malignancy within the last 5 years, except for carcinoma in situ of the cervix or non-melanoma skin cancer.
3. Previous chemotherapy for cancer or other malignant disease.
4. Charlson comorbidity index, excluding score for malignancy: (CCI) > 2, Comment: In patients 70-75 a CCI = 3 is allowed, see appendix B.
5. Inadequate organ function, suggested by the following laboratory results:

   a Absolute neutrophil count < 1,5 x 109/L

   b Platelet count < 100 x 109/L

   c Hemoglobin < 90 g/L

   d Total bilirubin greater than the upper limit of normal (ULN) unless the patient has documented Gilbert´s syndrome

   e ASAT (SGOT) and/or ALAT (SGPT) > 2,5 x ULN

   f ASAT (SGOT) and/or ALAT (SGPT) > 1,5 x ULN with concurrent serum alkaline phosphatase (ALP) > 2,5 x ULN

   g Serum creatinine clearance < 50 ml/min
6. Concurrent peripheral neuropathy of grade 3 or greater (NCI-CTCAE, Version 5.0).
7. Patient who is actively breast feeding.
8. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.
9. Patients with known deficiency of the DPD-enzyme who completely lack DPD.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Estimated)
Dates: Start 2019-12-20 (Actual); Primary Completion 2035-09 (Estimated); Study Completion 2035-09 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate. | Immediately after surgery
  Rate of pathological complete response, allowing residual dcis, at surgery after preoperative chemotherapy.
Primary translational outcome. | Immediately after surgery
  Pathological complete response rate, allowing residual dcis, stratified for homologous repair deficiency.

SECONDARY OUTCOMES:
Invasive Disease Free Survival (IDFS) | Throughout the study, an average of 3 years
  Invasive disease-free survival
Overall Survival (OS) | Throughout the study, an average of 5 years
  Overall survival
Breast Cancer Specific Survival (BCSS) | Throughout the study, an average of 3 years
  Breast cancer specific survival
Distant Recurrence Free Survival (DRFS) | Throughout the study, an average of 3 years
  Distant recurrence free survival.
Dose intensity | Immediately after surgery
  Actual dosis/dosis per protocol
Toxicity according to CTCAE version 5.0 | Immediately after surgery
  Rate of included patients with toxicity grade 3 or greater during study treatment

OTHER OUTCOMES:
Subset characterization (histological subtypes) | Immediately after surgery
  Distribution of different histopathological subsets of Triple Negative Breast Cancer (TNBC).
Subset characterization (germline mutations) | Immediately after surgery
  Distribution of subsets of Triple Negative Breast Cancer (TNBC) associated with different inherited breast cancer genes (BRCA1, BRCA2, PALB2, TP53, CHEK2, ATM, RAD51 C and RAD51D).
Subset characterization (somatic mutations) | Immediately after surgery
  Distribution of subsets of Triple Negative Breast Cancer (TNBC) associated with somatic mutations, (Eg BRCA1, BRCA2, PALB2, TP53, and other).
Subset characterization (epigenetic alterations) | Immediately after surgery
  Distribution of different subsets of Triple Negative Breast Cancer (TNBC) defined based on epigenetic alterations associated with silencing of BRCA1, RAD51 and related HRD-associated genes.
pCR and long term outcome in histologic subsets of TNBC | Immediately after surgery
  pCR rate in different histopathological subsets of Triple Negative Breast Cancer (TNBC).
pCR and long term outcome in subsets of TNBC defined based on occurrence of germline genetic alterations | Immediately after surgery
  pCR rate in subsets of Triple Negative Breast Cancer (TNBC) associated with different inherited breast cancer genes (BRCA1, BRCA2, PALB2, TP53, CHEK2, ATM, RAD51 C and RAD51D).
pCR and long term outcome in subsets of TNBC defined based on occurrence of somatic genetic alterations | Immediately after surgery
  pCR rate in subsets of Triple Negative Breast Cancer (TNBC) associated with somatic mutations, (Eg BRCA1, BRCA2, PALB2, TP53, and other).
pCR and long term outcome in subsets of TNBC defined on epigenetic alterations | Immediately after surgery
  pCR rate in different subsets of Triple Negative Breast Cancer (TNBC) based on epigenetic alterations associated with silencing of BRCA1, RAD51 and related HRD-associated genes.
pCR and long term outcome in immun marker defined subsets of TNBC | Immediately after surgery
  pCR rate in subsets of Triple Negative Breast Cancer (TNBC) associated with the expression of PDL1.

CONTACTS AND LOCATIONS:
Overall Officials: Niklas Loman, MD, PhD, Study Director — Lund University Hospital
Locations (24):
- Denmark (8):
  - Vejle Hospital, Vejle, Region Syd
  - Aalborg Universitetshospita, Aalborg
  - Rigshospitalet, Copenhagen
  - Sydvestjysk Sygehus, Esbjerg
  - Nordsjællands Hospital, Hillerød
  - Regionsjælland Næstved Sygehus, Næstved
  - Sønderborg sygehus, Sønderborg
  - Vejle syghus, Vejle
- Sweden (16):
  - Centralsjukhuset i Kristianstad, Kristianstad, Skåne County
  - Södra Älvsborgs Hospital, Borås
  - Gävle hospital, Department of Oncology, Gävle
  - Sahlgrenska University Hospital, Department of Oncology, Gothenburg
  - Halmstad Hospital, Department of Surgery, Halmstad
  - Ryhov Hospital, Jönköping
  - Karlstad Hospital, Karlstad
  - Skåne University Hospital, Department of Oncology, Malmo
  - Örebro University Hospital, Department of Oncology, Örebro
  - Capio S:t Göran Hospital, Department of Oncology, Stockholm
  - Södersjukhuset, Department of Oncology, Stockholm
  - Sundsvall hospital, Sundsvall
  - Norrland University Hospital, Department of Oncology, Umeå
  - Academical Hospital, Department of Oncology, Uppsala
  - Växjö Hospital, Department of Oncology, Vaxjo
  - Västmanlands Hopsital Västerås, Västerås

IPD SHARING:
Plan to Share IPD: No